CLINICAL TRIAL: NCT05330572
Title: Clinical and Molecular Correlates of Response to First Line Treatment in Lichen Planus
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-064-21
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Lichen Planus, Oral; Lichen Planus of Vulva
Keywords: oral lichen planus, vulvovaginal lichen planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Saliva
  * Oral mucosal swab
  * Venous blood sample
  * Vulvo-vaginal swab (where applicable)
  * Cervico-vaginal lavage (where applicable) All the above samples will be stored in media suitable for microbiological and immunological analysis. They will be either stored on ice for immediate processing or stored at -20° for the later analysis at the Institute of Medical Sciences, University of Aberdeen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral lichen planus: No interventions were administered to this group of patients as a part of the study.
  Interventions: Other: No interventions were administered to the patients as a part of this study.
- Oro-vulvovaginal lichen planus: No interventions were administered to this group of patients as a part of the study.
  Interventions: Other: No interventions were administered to the patients as a part of this study.

INTERVENTIONS:
Other: No interventions were administered to the patients as a part of this study. — No interventions were administered to the patients as a part of this study. Patients who were under topical steroid regime as a part of their management plan for lichen planus will be enrolled on the study. Details of prescribed topical steroid regime for lichen planus: type of corticosteroid, formulation, frequency of application, duration of treatment will be recorded.

SUMMARY:
Lichen planus is a common inflammatory (swelling and pain of tissue) disease in the general population that affects mostly the mouth although skin and genital areas can also be affected. It can cause considerable discomfort during activities such as eating, talking and tooth brushing and may impair sexual function with an overall deleterious impact on quality of life. There is also increased evidence of cancer in a subtype of lichen planus. Therefore, treatment is essential in these patients to control the symptoms and improve the quality of life.

Locally applied steroids are the first line medicines used in the treatment of patients with lichen planus. This medicine can only control the symptoms, but cannot cure the disease. In addition, this treatment cannot be effective in all patients with lichen planus. This may be attributed to differences in host factors, mouth bacteria and individual host responses to bacteria. The exact cause of this disease is also unknown. New studies have shown changes in the balance of mouth bacteria and host responses to bacteria in patients with lichen planus. So the main purpose of our study is to identify clinical(age, gender, related medical conditions, oral health and the presence of deleterious habits like smoking and alcohol consumption), molecular(analysis of oral microbes and immune markers) and histological factors (change within tissue) associated with poor response in lichen planus patients undergoing treatment with locally applied steroid medicines. Overall, knowledge of these factors associated with disease progression is sparse, which limits progress in the realm of development of novel and personalised treatment strategies. In this study, we explore the individual and combined role of different markers in lichen planus for improving diagnosis, predicting disease progression and treatment effectiveness.

DETAILED DESCRIPTION:
PARTICIPANT SELECTION AND ENROLMENT

IDENTIFYING PARTICIPANTS All participants will be selected from attendants of the Oral & Maxillofacial Unit, Women's Day Clinic and Aberdeen Dental School in the Foresterhill Campus. The research team will identify eligible participants for the study by screening through review of their electronic records. Caldicott Guardian approval will be sought for Sreedevi P.U to gain direct access to patient clinical records for screening purposes. Patients diagnosed with oral or oral and vulvovaginal lichen planus will be recruited into the study, only following biopsy confirmation. The diagnosis of lichen planus will be made on the basis of accepted clinical and histopathological findings, to meet the eligibility criteria, patients must be undergoing topical steroid therapy as a part of their management plan for lichen planus.

SCREENING FOR ELIGIBILITY Patients attending routine clinics will be screened for eligibility through review of their electronic records. Here, we emphasise that no study data will be recorded from participant's medical/dental records, until we have a written informed consent from them. Eligibility of patients will be checked for predefined inclusion/exclusion criteria by reviewing clinical and histopathological records of patients that have been diagnosed with lichen planus by the clinical research team.

CONSENTING PARTICIPANTS

Potentially eligible patients will be contacted through a research study information pack sent by post. The research study information pack will include: an invitation letter, a Patient Information Sheet (PIS), a return slip and pre-paid envelope for the patient to notify the research team of whether or not they wish to participate. If the patient is interested in taking part, they will be contacted by telephone by the research team to arrange a visit at a dedicated research study session. At this point, written informed consent will be obtained from potentially eligible patients after having a verbal discussion about the nature of the study and answering any questions the patient may have. Informed consent from patients with oral lichen planus will be obtained by Dr Sreedevi P.U and the research nurse named in this application will be involved in obtaining consent from patients with vulvovaginal disease. Patients will be consented for the following aspects:

1. Review of their medical and dental records
2. Analysis of the histological records associated with the lichen planus diagnosis
3. Provision of additional information relating to host factors potentially to lichen planus progression if not already available in the patient records.
4. Filling questionnaire related to stress levels.
5. Intraoral examination
6. Sample collection (blood, saliva, swabs)
7. Vulvovaginal examination and sampling (where relevant)
8. Follow-up post-treatment appointment.
9. Storage and use of their samples for ethically reviewed and approved future studies.
10. To be contacted by the study team for future ethically approved studies.

STUDY ASSESSMENTS

The following clinical information will be recorded for all patients if not already available through the patient's medical/dental records:

1. Dental/Medical History include past and current dental and medical conditions.
2. Social History include smoking status, alcohol consumption and stress levels. The 10-item Perceived Stress Scale (PSS-10) will be used to assess perceived stress level in the patients with lichen planus. It is a self-report scale which measures the degree to which situations over the last month in the respondent's life are appraised as unpredictable, uncontrollable and overloading.
3. Assessment of Oral Health

   Patients recruited for the study will undergo a partial assessment of oral health aimed at recording the following information:
   * Oral hygiene status To be assessed by performing Simplified Oral Hygiene Index (OHI-S) which has two components, the Debris Index-Simplified (DI-S) and the Calculus Index-Simplified (CI-S).
   * Basic periodontal examination A basic periodontal examination is a routine screening investigation carried out to assess periodontal health. It involves probing of the periodontal tissues to assess the presence of bleeding on probing, plaque and calculus deposits and the depth of any periodontal pockets which may be present. Basic periodontal examination will be conducted in accordance with the guidelines of the British Society of Periodontology.
   * Disease severity score of Lichen Planus It will be scored based on site of involvement, disease activity and pain using the best scoring system identified by conducting a systematic review.
   * Detail of prescribed topical steroid regime for lichen planus: type of corticosteroid, formulation, frequency of application, duration of treatment.
4. Vulvovaginal Examination Patients diagnosed with vulvo-vaginal lichen planus will undergo a vulval examination to formally score disease severity. A speculum examination will be performed to assess disease severity for those women with vaginal disease and to collect swab of vaginal secretions.
5. COLLECTION OF SAMPLES Samples (saliva, blood, oral swabs and vaginal sampling (where applicable) will be collected from the patient's who have started their topical steroid treatment, aimed at microbiome and immune markers analyses. Participants will need to undergo a second sampling after the completion of topical steroid treatment approximately two months after their first visit.

Saliva: For this study, we will collect two unstimulated whole saliva fasting samples, one sample for the study of inflammatory/immune factors, another sample for the microbiome studies. To reduce the number of variables that may interfere with composition of the microbial populations colonising the oral tissues, eligible patients will be asked not to use antibacterial mouthwashes for 48 hours prior to the visit. Patients will also be asked to preferably attend morning clinics so that samples can be collected before participants eat the breakfast.

Oral swabs: Two oral swabs (one from affected tissue, one from adjacent healthy tissue). Patients will be advised not to use antibacterial mouthwashes for 48 hours prior to the oral swabs. They will also be asked to attend the morning clinics to reduce the dietary influence on sampling results.

Vulvovaginal sampling: For all patients presenting with vaginal and/or vulval disease we will collect 1 cervico-vaginal lavage sample and up to 3 swabs representative of healthy and diseased areas. Participants will be asked to abstain from sex for 24 hours prior to their appointment.

Bloods: A blood sample (up to 40 ml) will also be collected from patients from whom baseline haematological and biochemical parameters (full blood count, haematinics, random blood glucose, liver function test and Urea &Electrolytes) are not available. An additional sample will also be collected for analysis of inflammatory markers.

All samples will be transferred to the Institute of Medical Sciences (University of Aberdeen) for microbiome and immune marker analysis.

Histological sections of biopsies conducted as part of routine clinical care will be sourced from the Grampian Biorepository for digital pathology studies.

DATA ANALYSIS Disease response after the completion of topical steroid treatment will be modelled using a linear regression model. The model will adjust for the baseline disease levels (measured using the lichen planus severity score) along with clinical and molecular characteristics and assess the relationship of these predictors with lichen planus severity after treatment. In the event that assumptions for the linear regression model on the observed data are not fulfilled, alternative modelling options such as ordinal regression or logistic regression model will be explored.

Microbial diversity will be assessed by molecular and microbial approaches including but not exclusively next-generation sequencing and multi-locus sequence typing. Analysis of data generated by next-generation sequencing will be carried out at the University of Aberdeen with reference made to the Human Oral Microbiome Database or the CORE database.

Analysis of host responses (including CD4+ helper and CD8+ cytotoxic T cells, their secreted pro-inflammatory and anti-inflammatory cytokine profiles, and any specific autoantibodies) will be carried out mainly by RT-PCR, immunoblotting and flow-cytometry.

Analysis of histopathological images will be aimed at recording the following information:

* Quantification of morphological parameters at the tissue and cellular levels
* Quantification of immune markers such as CD4+Tcells, Foxp3, CD8+T cells, PD-1, PDL-1 and TLRs.

The image processing and analysis will be conducted using the open access image analysis software packages ImageJ and QuPath.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years, with confirmed histopathological diagnosis of lichen planus and undergoing topical steroid therapy.
* Participants who have the capacity to consent.
* Participants who show a willingness to attend an initial appointment and a follow-up post-treatment appointment.

Exclusion Criteria:

* Patients on systemic steroids and other immunosuppressive agents for the treatment of lichen planus
* Cases of graft versus host disease or those suffering from other systemic inflammatory conditions mimicking lichen planus (e.g. connective tissue disease).
* Pregnant and lactating participants.
* Inability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be selected from attendants of the Oral & Maxillofacial Unit, Women's Day Clinic and Aberdeen Dental School in the Foresterhill Campus. Patients diagnosed with oral or vulvovaginal lichen planus will be recruited into the study, only following biopsy confirmation. The diagnosis of lichen planus will be made on the basis of accepted clinical and histopathological findings to meet the eligibility criteria. Patients who have been advised to use topical steroid therapy as a part of their management plan for lichen planus.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification of host related factors associated with poor response to topical steroid therapy in patients with lichen planus. | change in disease severity score of lichen planus from baseline (start of topical steroid treatment) to completion of topical steroid therapy( 2 months after the first visit)
  Correlation between the host related factors (clinical factors) and change from baseline in lichen planus disease severity score at 2 months will be assessed.
Identification of inflammatory/immune markers associated with poor response to topical steroid therapy in patients with lichen planus. | change in disease severity score of lichen planus from baseline (start of topical steroid treatment) to completion of topical steroid therapy( 2 months after the first visit)
  Correlation between the inflammatory/immune markers in saliva or serum and change from baseline in lichen planus disease severity score at 2 months will be assessed.
Determination of microbiome characteristics predictive of response to treatment. | change in disease severity score of lichen planus from baseline (start of topical steroid treatment) to completion of topical steroid therapy( 2 months after the first visit)
  Correlation between oral microbiota and change from baseline in lichen planus disease severity score at 2 months will be assessed.
Identification of histopathological morphological markers associated with poor response to topical steroid therapy in patients with lichen planus. | change in disease severity score of lichen planus from baseline (start of topical steroid treatment) to completion of topical steroid therapy( 2 months after the first visit)
  Quantification of histopathological morphological markers will be determined by analysing histopathological images of oral lichen planus using software applications ImageJ and QuPath. Correlation between these factors and change from baseline in lichen planus disease severity score at 2 months will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Karolin Hijazi, Principal Investigator — University of Aberdeen
Locations (2):
- United Kingdom (2):
  - University of Aberdeen, Aberdeen, Aberdeen, Scotland
  - Aberdeen Dental School, Aberdeen

IPD SHARING:
Plan to Share IPD: No